CLINICAL TRIAL: NCT00241228
Title: Impact of High-volume Veno-venous Continuous Hemofiltration in the Early Management of Septic Shock Patients With Acute Renal Failure
Brief Title: Haemofiltration Study : IVOIRE (hIgh VOlume in Intensive Care)
Acronym: IVOIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9410-04; 2004-024
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Shock, Septic; Renal Failure, Acute
Keywords: Shock, Septic; Renal Failure, Acute; Venovenous Hemofiltration; Randomized Controlled Trial; Multicenter Study; Mortality
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury | interventions — Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Volume (Experimental): ultra filtration : High volume : 70 ml/kg/h
  Interventions: Device: Venovenous haemofiltration (renal replacement therapy)
- Medium Volume (Active Comparator): Ultra filtration : conventional volume : 35 ml/kg/h
  Interventions: Device: Venovenous haemofiltration (renal replacement therapy)

INTERVENTIONS:
Device: Venovenous haemofiltration (renal replacement therapy) — High Volume ultra filtration (70 ml/kg/h)
  Arms: High Volume
Device: Venovenous haemofiltration (renal replacement therapy) — Conventional Volume (35 ml/kg/h)
  Arms: Medium Volume

SUMMARY:
Sepsis and septic shock are still important causes of mortality in intensive care medicine. Renal replacement therapy by standard volume haemofiltration is currently used, but a higher-volume haemofiltration may improve the prognosis. The study is a prospective randomized multicenter trial comparing two treatments in patients suffering from septic shock complicated with acute renal failure admitted to ICU. One group will be treated by early high volume haemofiltration (70 ml/kg/h) and the second group by standard volume haemofiltration (35 ml/kg/h). The main outcome will be one-month mortality.

DETAILED DESCRIPTION:
Background

Sepsis and septic shock are still important causes of mortality in intensive care medicine nowadays. Mortality ranges from 40 up to 80 % depending on the number of organ failures. Therapeutic strategy consists of two major components: haemodynamic stabilization with restoration of adequate arterial pressure and optimization of peripheral perfusion delivery, and infection treatment. Mortality remains high despite the use of new antimicrobial therapy and adjuvant therapies such as activated protein C, low dose corticoids and haemofiltration. Initial observations in patients with acute renal failure treated by haemofiltration showed azotemia control, restoration of the sodium-water balance, elimination of inflammatory mediators and improvement of the cardiac and pulmonary functions was demonstrated independently of a negative water balance. There is no human randomized study so far demonstrating these preliminary findings. Nevertheless, several authors have demonstrated inflammatory mediators elimination by the use of haemofiltration. Moreover, the clinical improvement seems to be related to the ultra filtration dose and to the early initiation of therapy. Joannes-Boyau et al carried out a pilot study in abdominal surgery patients demonstrating that the use of high volume haemofiltration in patients with septic shock and multiple organ failure restores hemodynamic stability with drastic reductions in catecholamine requirements and a substantial reduction of observed vs. expected mortality.

Objectives

The principal objective of the study is to evaluate the effect of early Continuous High Volume Haemofiltration on 28-day mortality in patients with septic shock complicated by acute renal failure. The secondary objectives are to assess the effect of High Volume Haemofiltration on haemodynamics, doses of catecholamines, organ failures, duration of mechanical ventilation, duration of renal replacement therapy need, morbidity, length of ICU and hospital stay, and 60- and 90-day mortality.

Study design

Open label randomized multicenter controlled trial on two parallel groups of patients with septic shock and acute renal failure admitted to ICU, treated early either by high volume (70 ml/kg/h) or by standard volume (35 ml/kg/h) haemofiltration.

Eligibility criteria

Inclusion criteria. Septic shock (Bone criteria) for less than 24 hours, RIFLE criteria : injury or worse, age over 18 years, and written informed consent by next of kin. Non inclusion criteria. Cirrhosis, age over 80 years, life expectancy less than 3 months or metastatic cancer.

Intervention

High volume (70 ml/kg/h) vs. standard volume (35 ml/kg/h) haemofiltration during 96 hours. Further renal replacement therapy (if haemofiltration, only standard volume is allowed) may be used according to investigator decision.

Primary endpoint

All cause 28-day mortality.

Statistical aspects

460 patients are planned to be included (230 in each group). A 15 % absolute reduction in 28-days all-cause mortality in the high volume group compared with the standard group is expected. However, as this reduction might be greater, an interim analysis is planned when half of the total sample size will have been included. Data will be analyzed on an intention-to-treat basis.

Duration of the study: 3 years.

ELIGIBILITY:
Inclusion Criteria:

* septic shock (Bone criteria) for less than 24 hours
* RIFLE criteria : injury or worse
* age over 18 years
* written informed consent by next of kin.

Exclusion Criteria:

* cirrhosis
* age over 80 years
* life expectancy less than 3 months or metastatic cancer
* for women : pregnancy and breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
all-cause mortality. | 28-day

SECONDARY OUTCOMES:
Haemodynamic parameters and volume loading | Every 12 hours during 96 hours after inclusion
Doses and duration of catecholamine infusions | Every 12 hours during 96 hours after inclusion
Organ failures | During 96 hours after inclusion
Duration of mechanical ventilation | Total during the stay in intensive care
Duration of renal replacement therapy | Total during the stay in Intensive Care Unity (ICU)
Morbidity | Total during the stay in intensive care
Length of stay in ICU and hospital | End of hospitalization
Mortality | in ICU (96 first hours after inclusion), 60 and 90-day

CONTACTS AND LOCATIONS:
Overall Officials: Olivier JOANNES-BOYAU, Dr, Principal Investigator — University Hospital, Bordeaux, France; Patrick HONORE, Dr, Principal Investigator — Quuen Astrid Military Hospital, BRUXELLES - Belgium; Paul Perez, Dr, Study Chair — University Hospital, Bordeaux, France
Locations (16):
- Belgium (5):
  - Cliniques de l'Europe, Brussels
  - Astrid Queen Military Hospital, Bruxelles (Neder Over Hembeek)
  - TIVOLI Hospital, La Louvière
  - University Hospital, Liège
  - St-Pierre Para-University Hospital, Ottignies-Louvain-la-Neuve
- France (9):
  - Hospital, Agen
  - Clinic Bordeaux Nord, Bordeaux
  - University Hospital, Brest
  - University Hospital, Grenoble
  - Hospital R Boulin - Libourne, Libourne
  - University Hospital, Lyon
  - Aphp - Hegp, Paris
  - Service d'Anesthésie-Réanimation II, Groupe Hospitalier Sud, CHU de Bordeaux, Pessac
  - Hospital, Tourcoing
- Netherlands (2):
  - Hospital, Delf
  - Hospital, Heerlen

REFERENCES:
- [Derived] Medica D, Quercia AD, Marengo M, Fanelli V, Castellano G, Fabbrini P, Migliori M, Merlotti G, Camussi G, Joannes-Boyau O, Honore PM, Cantaluppi V. High-volume hemofiltration does not protect human kidney endothelial and tubular epithelial cells from septic plasma-induced injury. Sci Rep. 2024 Aug 7;14(1):18323. doi: 10.1038/s41598-024-69202-z. PMID 39112634
- [Derived] Joannes-Boyau O, Honore PM, Perez P, Bagshaw SM, Grand H, Canivet JL, Dewitte A, Flamens C, Pujol W, Grandoulier AS, Fleureau C, Jacobs R, Broux C, Floch H, Branchard O, Franck S, Roze H, Collin V, Boer W, Calderon J, Gauche B, Spapen HD, Janvier G, Ouattara A. High-volume versus standard-volume haemofiltration for septic shock patients with acute kidney injury (IVOIRE study): a multicentre randomized controlled trial. Intensive Care Med. 2013 Sep;39(9):1535-46. doi: 10.1007/s00134-013-2967-z. Epub 2013 Jun 6. PMID 23740278